CLINICAL TRIAL: NCT00376636
Title: A Phase IIa, Double-Blind, Placebo-Controlled, Randomised, Parallel-Design, Four-Week Study to Investigate the Safety and Efficacy of the Oral Renin Inhibitor SPP635 Once Daily in Patients With Mild to Moderate Hypertension
Brief Title: Phase IIa Safety and Efficacy Study of SPP635 in Mild to Moderate Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Speedel Pharma Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPP635CRD04
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2007-10-30 (Estimated); Status verified 2006-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SPP635 (drug)

SUMMARY:
This study is conducted to investigate the effect of the oral renin inhibitor SPP635 on blood pressure in patients with mild to moderate hypertension.

DETAILED DESCRIPTION:
Renin-Angiotensin system blockade is a well established target for treatment of high blood pressure. Blocking the system at the initial step, however, is a rather new concept that could only be implemented very recently through the availability of novel, oral, renin inhibitors. This study investigates the safety and efficacy of a novel oral renin inhibitor, SPP635.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients with mild to moderate hypertension

Exclusion Criteria:

* female patients of child-bearing potential or breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-10; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Lowering of systolic office blood pressure | four weeks
Lowering of diastolic office blood pressure | four weeks

SECONDARY OUTCOMES:
Lowering of systolic and diastolic blood pressure (ABPM) | four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sybille Baumann-Noss, MD, Principal Investigator — IKP Bobenheim GmbH
Locations (1):
- IKP Bobenheim GmbH, Mannheim, Germany